CLINICAL TRIAL: NCT02121366
Title: Endoscopic Ultrasound (EUS)-Guided Ethanol Ablation of an Insulinoma - A Multi-center Prospective Cohort Study
Brief Title: EUS-guided Ethanol Ablation of an Insulinoma
Acronym: EUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Shanyu Qin, First Affiliated Hospital of Guangxi Medical University, Guangxi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUS0511
Record Dates: First submitted 2014-03-26; First posted 2014-04-23 (Estimated); Last update posted 2014-04-23 (Estimated); Status verified 2014-04

CONDITIONS: Insulinoma
Keywords: Endoscopic Ultrasound-Guided Fine Needle Aspiration; Insulinoma; Ethanol; Ablation Techniques
MeSH Terms: conditions — Insulinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Insulinoma (Experimental): Patients with Insulinomas will received EUS-guided ethanol ablation therapy
  Interventions: Procedure: EUS-guided ethanol ablation

INTERVENTIONS:
Procedure: EUS-guided ethanol ablation — Diagnostic evaluation for suspected insulinoma is performed by cytology or immunohistochemistry. EUS-FNA is performed to obtain samples. After puncturing with the needle, ethanol under the guidance of EUS was injected into the lesion. The amount of ethanol is administrated according to the size of lesion.

SUMMARY:
The present study aims to evaluate the feasibility, safety and efficacy of EUS-guided ethanol ablation of an insulinoma.

DETAILED DESCRIPTION:
As the major insulinomas are functioning islet cell tumors, surgical resection is currently first-line therapy for or treatment of insulinomas. However, the surgical resection of pancreatic neoplasm is conditional for specific patients and may be associated with substantial life-threatening complications. Several studies declared that endoscopic ultrasound (EUS)-guided lavage may offer an alternative to surgical resection of insulinomas. Nevertheless, their sample sizes were small and conclusions were built based on short-term outcomes. In addition, the amount of ethanol administrated for different types of insulinomas were inconsistent among those studies.

The present study aims to evaluate the safety, feasibility and efficacy of EUS-guided ethanol ablation therapy of insulinomas. We will use cytopathology and immunohistochemistry in combination with EUS-FNA for diagnosis of insulinoma. After EUS-guided ethanol ablation therapy, the safety and efficacy will be assessed at the baseline and different time points during follow-up by physicians blinded to the treatment or control status.

ELIGIBILITY:
Inclusion Criteria:

1. Adults: at least 18 years.
2. Patients with insulinomas which are evaluated by histopathology .
3. patients who have signed a written consent form.

Exclusion Criteria:

1. Patients whose condition is not suitable for the endoscopic procedure.
2. Patients who have blood coagulation dysfunction.
3. Patients who have mental disorders.
4. Patients who have mild or severe cardiorespiratory insufficiency.
5. Patients who have hypertension and could not be controlled to safe level.
6. Pregnant and lactating women.
7. Patients whose conditions are not suitable for the present study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy of EUS-guided ethanol ablation | 1 to 12 month
  Volumes of insulinomas before and after treatment, which are measured by cross-sectional imaging test (CT or MRS).
Safety of EUS-guided ethanol ablation | 1 to 12 month
  Number of subjects with post-procedure adverse events

SECONDARY OUTCOMES:
Technical feasibility | during the procedure of treatment
  Technical success was defined as ethanol is injected and lavaged into target tissue.

CONTACTS AND LOCATIONS:
Overall Officials: Shanyu Qin, MD. Ph.D., Study Chair — First Affiliated Hospital of Guangxi Medical University
Locations (1):
- First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi, China